CLINICAL TRIAL: NCT00319176
Title: Evaluation of Pre-dose and Post-dose Anti-factor Xa Levels With Enoxaparin Use During Pregnancy
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Long Beach Memorial Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 162-04
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Pregnancy
Keywords: Pregnancy; Enoxaparin; Anticoagulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Venous thromboembolism is a condition that causes formation of blood clots in the body. It may have life threatening consequences if the leg veins, lungs or the brain blood vessels are involved. In pregnancy, a woman's baseline risk for forming blood clots is increased.

Women with a known prior blood clot during pregnancy, artificial heart valves or other genetic conditions are at a very high risk for these complications during their pregnancy. It has been well established that these women benefit from medical treatment with a blood thinning medication in their pregnancies to prevent further formation of blood clots. These medications are called Heparins and are given as shots. Prior studies have suggested that a type of Heparin called "low molecular weight heparin" (Enoxaparin=Lovenox®) is well suited for use in pregnancy as it does not affect the baby and has a very low complication rate.

The standard dose given for treatment of these patients has been established previously. However, there is a concern that complications may occur if the concentration of this medication falls below its effective level. It is of particular importance in pregnancy, as the rate of breakdown of this medication increases in pregnancy and may lead to lowering of its effective levels.

Our study will evaluate the blood levels of enoxaparin before and after administration of this medication in pregnant women who are receiving this drug for treatment. This will determine whether an increase in the dose or an increase in the frequency of dosing might further improve the standard of care.

DETAILED DESCRIPTION:
Study Design This is a prospective, non-blinded, pilot study of gravid patients receiving treatment doses of enoxaparin therapy.

Subjects Subjects will include pregnant women at all gestational ages already receiving a treatment (therapeutic) dose regimen of enoxaparin (1 mg/kg ± 20% SC BID). Patients who are managed by one of the principal or co-investigators at Long Beach Memorial Medical Center Women's Hospital may be readily identified as potential candidates for the study. Additionally, other perinatologists, obstetricians, and resident physicians who prescribe enoxaparin for their patients may ask a co-investigator to consent a woman for the study. Women will be individually counseled by their physicians as to the best antithrombotic drug therapy to use during pregnancy, and in the case of enoxaparin use, may be asked to participate in this study.

Inclusion Criteria:

1. Nulliparous or multiparous women with intrauterine pregnancies who are receiving twice daily treatment doses of enoxaparin (1 mg/kg ± 20% SC BID).
2. Subjects who consent to the study.

Exclusion Criteria:

1. Women who are not pregnant.
2. Women who are receiving enoxaparin at prophylactic doses (i.e., 30 mg twice daily or 40 mg daily).
3. Women who are currently receiving another LMWH or UFH.
4. Women who are receiving other concomitant anticoagulant medications, such as warfarin, lepirudin, or argatroban.
5. Subjects who are unable or unwilling to give informed consent.
6. Women who, in the judgment of the investigators, would not be in the best interest of the patient to participate in the study.

Methods Women who are eligible and consent to participate in the study will receive the twice daily standard enoxaparin dose, as prescribed by her physician. Enoxaparin (Lovenox®; Aventis Pharmaceuticals) will be filled by the hospital's inpatient pharmacy department at Long Beach Memorial Medical Center, as long as the subject is admitted to the hospital.

If the patient is an inpatient, the patient's nurse will administer the doses as per hospital drug administration policy, subcutaneously at 8:00 am and 8:00 pm. Immediately prior to receiving her fourth dose, an anti-factor Xa level will be drawn - called the "pre-dose" level. Waiting until this time period allows enoxaparin to reach adequate steady-state levels based on an average elimination half-life of 4.5 hours (range 3 to 6 hours). Three hours after the fourth dose of enoxaparin is administered, another anti-factor Xa level will be drawn - called the "3-hour post-dose" level. Eight hours after the fourth dose of enoxaparin is administered, an anti-factor Xa level will be drawn as well - called the "8-hour post-dose" level. The same set of levels will be measured during admission after any dosage adjustments. Enoxaparin dosage changes will be made at the discretion of the treating physician.

If the patient is an outpatient, she will be instructed to adjust her medication administration times so that the timing of her pre-dose, 3-hour post-dose, and 8-hour post-dose levels fall within the day's working hours. We will also ensure that the drug is at steady state prior to obtaining the blood samples by verifying that she has had at least 3 doses of the medication.

Blood obtained for lab draws are centrifuged for 15 minutes at a speed of 3,000 g, and at a temperature of around 18ºC. Centrifugation is performed within 1 hour after sample collection. The plasma samples are then analyzed in batches for anti-factor Xa activity by amidolytic assay, done at noon daily in Long Beach Memorial's Department of Pathology (Coagulation). If the assay is not performed within 30 minutes of centrifugation, the plasma is frozen. Plasma samples may be frozen for up to 6 months. The minimum detectable limit of this assay is 0.1 U/ml, and the linearity range extends to 2.0 U/ml. Therapeutic anti-factor Xa activity is designated as 0.5-1.2 U/ml. The coefficient of variation for this assay is 98%.13

Statistical Analysis:

The plasma anti-factor Xa activity levels measured for this study will be analyzed by comparing the incidence of pre-dose and post-dose levels that fall in the therapeutic anti-factor Xa activity range. The incidence of therapeutic and non-therapeutic anti-factor Xa post-dose levels will be compared to pre-dose levels using Student's t-test and Fisher's exact. If dose adjustments are necessary, changes will be made using the traditional method of post-dose level analysis. Mean time to anti-factor Xa therapeutic range will be evaluated as well.

Subjects will be treated in this study in an intent-to-treat basis, and data will be analyzed as such. Anticoagulation therapy postpartum will be decided at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous or multiparous women with intrauterine pregnancies who are receiving twice daily treatment doses of enoxaparin (1 mg/kg ± 20% SC BID).
2. Subjects who consent to the study.

Exclusion Criteria:

1. Women who are not pregnant.
2. Women who are receiving enoxaparin at prophylactic doses (i.e., 30 mg twice daily or 40 mg daily).
3. Women who are currently receiving another LMWH or UFH.
4. Women who are receiving other concomitant anticoagulant medications, such as warfarin, lepirudin, or argatroban.
5. Subjects who are unable or unwilling to give informed consent.
6. Women who, in the judgment of the investigators, would not be in the best interest of the patient to participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obstetrics clinic
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2004-04; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afshan B Hameed, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States

REFERENCES:
- [Derived] Friedrich E, Hameed AB. Fluctuations in anti-factor Xa levels with therapeutic enoxaparin anticoagulation in pregnancy. J Perinatol. 2010 Apr;30(4):253-7. doi: 10.1038/jp.2009.164. Epub 2009 Oct 15. PMID 19829297